CLINICAL TRIAL: NCT05224895
Title: Evaluation of the Effect of Trendelenburg Position on the Ultrasonographic Airway Measurements and Critical Respiratory Events
Brief Title: The Effect of Trendelenburg Position on the Ultrasonographic Airway Measurements
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, ismail aytaç, principal investigator, Ankara City Hospital Bilkent
Other Study IDs: E1-21-2231
Record Dates: First submitted 2021-12-26; First posted 2022-02-04 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Airway Edema; Ultrasonography; Robotic Surgical Procedures; Postoperative Respiratory Complication
Keywords: Airway edema; ultrasonography; Robotic surgical procedures; Postoperative Respiratory Complication
MeSH Terms: interventions — Anesthesia, General; Head-Down Tilt

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General Anesthesia in Trendelenburg position for robotic prostatectomy
  Interventions: Procedure: General Anesthesia in Trendelenburg position for robotic prostatectomy

INTERVENTIONS:
Procedure: General Anesthesia in Trendelenburg position for robotic prostatectomy — in this arm, changes in preoperative and postoperative airway measurements and correlation with postoperative critical airway events will be monitored.

SUMMARY:
The aim of this study is to compare the changes in upper airway edema with the preoperative and postoperative ultrasonographic measurements of patients who undergo pobotic prostatectomy in the trendelenburg position.

The secondary aim is to investigate the correlation between OSAS risk levels determined by the STOP-BANG score in the preoperative period of the patients participating in the study airway ultrasound measurements and postoperative critical respiratory events in the preoperative and postoperative period.

DETAILED DESCRIPTION:
In the preoperative period, age, body weight, height, neck circumference, comorbidities (Charlson comorbidity index), ASA score, Modified mallampati classification, STOP-BANG risk score will be recorded.Intraoperative monitorization data will be recorded.

Following ultrasonographic airway measurements will be performed preoperatively and postoperatively.

A low frequency convex probe will be used for ultrasonography. To achieve a fixed position of the tongue, patients will be placed supine without a pillow, with their head fully tilted back, and asked to hold their tongue loosely, without phonation, with their mouth closed and tongue tips lightly touching the incisors. The probe will be placed under the chin in the median sagittal plane and adjusted to obtain a clear median sagittal tongue view.

Tongue thickness: When the ultrasound probe is placed under the chin on the median sagittal plane, with the mouth closed in the supine position, the tongue is in a natural position and the patient is silent, and the tongue root is displayed on the screen, the maximal vertical diameter from the tongue surface to the submental skin will be measured and recorded as tongue thickness .

Median sagittal tongue cross-sectional area: The sagittal cross-sectional area of the tongue will then be measured by tracing the circumference of the tongue on the ultrasound machine.

Tongue width: The tongue width will then be obtained by measuring the distance between the probe placed transversely under the chin and the furthest points in the middle of the tongue in order to obtain as complete a tongue contour as possible.

Tongue volume: Tongue volume will then be obtained by multiplying the mid-sagittal tongue cross-sectional area by the tongue width, as described in previous studies .

Lateral parapharyngeal wall thickness: The lateral parapharyngeal wall thickness will be measured with a linear probe placed laterally into the cervical region in the direction of the external auditory canal to visualize the branching of the carotid artery. The lateral edge of the pharynx will be visualized as a hyperechoic line. Vibration artifacts and pharyngeal position will be confirmed by swallowing the patient. The distance between the arteria carotid interna and the echogenic surface of the pharynx and the distance between the skin and the lateral wall of the pharynx will be measured .

Patients will be monitorized for critical respiratory events (CRE) postoperatively A PACU CRE is defined as, any unexpected hypoxemia (hemoglobin oxygen saturation < 90%), hypoventilation (respiratory rate < 8 bpm or arterial carbon dioxide tension > 50 mmHg), or upper airway obstruction (stridor or laryngospasm) will be considered as requiring active and specific intervention (ventilation, tracheal intubation, opioid or muscle relaxant antagonism, oral/nasal airway or airway manipulation).

1. Upper airway obstruction requiring intervention (jaw thrust, oral airway);
2. Mild to moderate hypoxemia (SpO2=93%-90%) that does not improve after active interventions in 3 L nasal cannula oxygen (increasing O2 flows to >3 L/min, high-flow surface application mask O2, verbal requests to breathe deeply, tactile stimulation);
3. Severe hypoxemia (SpO2<90%) on 3 L nasal cannula O2, hypoxemia that does not improve after treatment (increased O2 flows >3 L/min, high-flow face mask O2 application, verbal requests deep breathing, tactile stimulation);
4. Respiratory distress or signs of impending respiratory failure (respiratory rate >20/min, use of accessory muscles, tracheal tugging);
5. Inability to take deep breaths when requested by the PACU nurse;
6. The patient complains of symptoms of respiratory or upper airway muscle weakness (difficulty breathing, swallowing or speaking);
7. Patient requiring reintubation in the PACU;
8. Clinical evidence or suspected pulmonary aspiration after tracheal extubation (gastric contents and hypoxemia observed in the oropharynx)

ELIGIBILITY:
Inclusion Criteria:

1. Robotic Laparoscopic Prostatectomy
2. ASA I-II-III-IV risk group -

Exclusion Criteria:

1. contraindication of trendelenburg position,
2. history of maxillofacial deformity, tumor or trauma,
3. history of difficult airway,
4. decompensated cardiac, respiratory, hepatic, renal disease,
5. with cervical spine fracture
6. patient refusal -

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participants who undergo robotic prostatectomy in Ankara City Hospital
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Preoperative Tongue thickness | Baseline, preoperative
  When the ultrasound probe is placed under the chin on the median sagittal plane, with the mouth closed in the supine position, the tongue is in a natural position and the patient is silent, and the tongue root is displayed on the screen, the maximal vertical diameter from the tongue surface to the submental skin will be measured and recorded as tongue thickness
postoperative Tongue thickness1 | immediately postextubation
  When the ultrasound probe is placed under the chin on the median sagittal plane, with the mouth closed in the supine position, the tongue is in a natural position and the patient is silent, and the tongue root is displayed on the screen, the maximal vertical diameter from the tongue surface to the submental skin will be measured and recorded as tongue thickness
postoperative Tongue thickness2 | postoperative 2. hour
  When the ultrasound probe is placed under the chin on the median sagittal plane, with the mouth closed in the supine position, the tongue is in a natural position and the patient is silent, and the tongue root is displayed on the screen, the maximal vertical diameter from the tongue surface to the submental skin will be measured and recorded as tongue thickness
preoperative Tongue volume | Baseline, preoperative
  Tongue volume will then be obtained by multiplying the mid-sagittal tongue cross-sectional area by the tongue width
postoperative Tongue volume1 | immediately postextubation
  Tongue volume will then be obtained by multiplying the mid-sagittal tongue cross-sectional area by the tongue width
postoperativeTongue volume2 | postoperative 2. hour
  Tongue volume will then be obtained by multiplying the mid-sagittal tongue cross-sectional area by the tongue width
Preoperative Lateral parapharyngeal wall thickness | Baseline, preoperative
  The distance between the arteria carotid interna and the echogenic surface of the pharynx and the distance between the skin and the lateral wall of the pharynx will be measured
postoperative Lateral parapharyngeal wall thickness1 | immediately postextubation
  The distance between the arteria carotid interna and the echogenic surface of the pharynx and the distance between the skin and the lateral wall of the pharynx will be measured
postoperative Lateral parapharyngeal wall thickness2 | postoperative 2. hour
  The distance between the arteria carotid interna and the echogenic surface of the pharynx and the distance between the skin and the lateral wall of the pharynx will be measured
Number of participants with Critical respiratory events | Within postoperative 2 hours
  A PACU critical respiratory event (CRE), any unexpected hypoxemia (hemoglobin oxygen saturation < 90%), hypoventilation (respiratory rate < 8 bpm or arterial carbon dioxide tension > 50 mmHg), or upper airway obstruction (stridor or laryngospasm) will be considered as requiring active and specific intervention (ventilation, tracheal intubation, opioid or muscle relaxant antagonism, oral/nasal airway or airway manipulation).

CONTACTS AND LOCATIONS:
Overall Officials: betül güven aytaç, Principal Investigator — ankara ch bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided